CLINICAL TRIAL: NCT04096248
Title: Non-Contrast CT vs CTP or MRI Selection vs Medical Management in Late Presentation of Large Vessel Occlusion Stroke, 6-24 Hours. A Multicenter Retrospective Study
Brief Title: CT (Computerized Tomography) for Late EndovasculAr Reperfusion
Acronym: CLEAR
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Collaborators: Medtronic (Industry); Society of Vascular and Interventional Neurology (Unknown)
Responsible Party: Sponsor
Other Study IDs: H-37843
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Stroke, Cardiovascular
Keywords: Large vessel occlusion; CT [Computed Tomography]; CTP [Computed Tomography (CT) Perfusion]; Modified Rankin score; ASPECTS (Alberta Stroke Program Early CT Score)
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this multicenter, retrospective, cross-sectional, chart review study is to compare outcomes (disability, complications and mortality) of patients with large vessel occlusion stroke presenting at late time window selected by either Non-Contrast CT (NCCT) only, advanced imaging with CTP (Computed Tomography Perfusion), MRI (Magnetic Resonance Imaging), or medical management.

Boston Medical Center (BMC) will serve as the main data coordinating site. Fifteen additional sites will seek local IRB approval or ethics approval. The aggregated de-identified data will be analyzed comparing types of interventions and outcomes by type of imaging or medical management.

DETAILED DESCRIPTION:
Additional subgroup analysis that are planned include:

1. Futile Reperfusion in the Extended Window.

   We will evaluate clinical, imaging and time metric factors associated with successful reperfusion yet poor outcomes (modified Rankin 3-6) in the 6-24 hour window.

   An evaluation of factors associated with symptomatic intracranial hemorrhage and mortality will be conducted.
2. Pre-Stroke disability.

   1. EVT patients treated in the extended window compared to Medical Management
   2. EVT patients treated in the extended window with pre-existing disability vs. those without pre-existing disability
3. Intravenous Thrombolysis in the Extended Window

   We aim to compare the safety and outcomes of bridging IVT in patients with acute ischemic stroke due to large vessel occlusion (LVO) who underwent EVT 6 to 24 hours after time-last-known-well.
4. Medical Management vs CT selected Patients

   We hypothesize that in patients with large vessel occlusion in the anterior circulation presenting in the 6 to 24 hour window, patients who are selected by non-contrast CT and treated with endovascular therapy have more favorable outcomes (ordinal mRS shift) as compared to patients who are medically managed.
5. Sex differences in the Extended Window

   In this study we aim to asses whether there are sex differences in clinical outcomes and safety of EVT in patients presenting in the 6-24 hour time window.
6. Transfer Analysis

It is not well established whether transfer patients presenting in the extended window should have repeat imaging upon receipt at the endovascular center after an interim time window.

We hypothesize that within a 0 to 2, or 2 to 4 hour delay between images of the primary stroke center to receiving endovascular center, transferred patients in the extended window, who undergo thrombectomy with successful reperfusion will have similar outcomes in patients with or without repeat imaging at the receiving center.

We aim to compare the safety and outcomes of late-window bridging IVT vs. direct EVT for LVO acute ischemic stroke in the 6-24 hour time window.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting 6-24 hours from last known well with large vessel occlusion stroke
* ASPECTS score 5 or greater from last known well
* January 1, 2014 to May 1, 2022

Exclusion Criteria:

-Time last seen well to treatment <6 hours from last known well

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective chart abstraction will be done on consecutive patients treated with a large vessel occlusion stroke who meet the inclusion and none of the exclusion criteria between January 1, 2014 and May 1, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 2790 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2021-05-23 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Change in patients' disability based on a Modified Rankin Scale | baseline, 90 days
  The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 5. Lower scores correlate with less disability/dependence.

SECONDARY OUTCOMES:
Intracranial hemorrhage incidence | 90 days
  Number of cases of intracranial hemorrhage divided by appropriate denominator.
Mortality rate | 90 days
  Number of deaths divided by appropriate denominator.

CONTACTS AND LOCATIONS:
Overall Officials: Thanh Nguyen, MD, Principal Investigator — Boston Medical Center
Locations (19):
- United States (7):
  - Grady Health; Marcus Stroke & Neuroscience Center, Atlanta, Georgia
  - Boston Medical Center, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Cooper University Health Care, Camden, New Jersey
  - Upstate University Hospital, Syracuse, New York
  - University of Toledo, Toledo, Ohio
  - Mercy Health Neuroscience Institute, Toledo, Ohio
- UZ Leuven, Leuven, Belgium
- Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec, Canada
- Helsinki University Hospital, Helsinki, Finland
- Universite de Lille, Lille, France
- Germany (2):
  - University Hospital Carl Gustav Carus, Dresden
  - Heidelberg University, Heidelberg
- Japan (2):
  - National Cerebral and Cardiovascular Center, Osaka
  - National Hospital Organization Osaka National Hospital, Osaka
- Hospital de Egas Moniz, Lisbon, Portugal
- Val D'Hebron, Barcelona, Spain
- Switzerland (2):
  - Bern University Hospital, Bern
  - Lausanne University Hospital, Lausanne

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Nguyen TN, Abdalkader M, Nagel S, Qureshi MM, Ribo M, Caparros F, Haussen DC, Mohammaden MH, Sheth SA, Ortega-Gutierrez S, Siegler JE, Zaidi S, Olive-Gadea M, Henon H, Mohlenbruch MA, Castonguay AC, Nannoni S, Kaesmacher J, Puri AS, Seker F, Farooqui M, Salazar-Marioni S, Kuhn AL, Kaliaev A, Farzin B, Boisseau W, Masoud HE, Lopez CY, Rana A, Kareem SA, Sathya A, Klein P, Kassem MW, Ringleb PA, Cordonnier C, Gralla J, Fischer U, Michel P, Jovin TG, Raymond J, Zaidat OO, Nogueira RG. Noncontrast Computed Tomography vs Computed Tomography Perfusion or Magnetic Resonance Imaging Selection in Late Presentation of Stroke With Large-Vessel Occlusion. JAMA Neurol. 2022 Jan 1;79(1):22-31. doi: 10.1001/jamaneurol.2021.4082. PMID 34747975
- [Result] Seker F, Qureshi MM, Mohlenbruch MA, Nogueira RG, Abdalkader M, Ribo M, Caparros F, Haussen DC, Mohammaden MH, Sheth SA, Ortega-Gutierrez S, Siegler JE, Zaidi SF, Olive-Gadea M, Henon H, Castonguay AC, Nannoni S, Kaesmacher J, Puri AS, Farooqui M, Salazar-Marioni S, Kuhn AL, Kiley NL, Farzin B, Boisseau W, Masoud HE, Lopez CY, Rana A, Abdul Kareem S, Sathya A, Klein P, Kassem MW, Cordonnier C, Gralla J, Fischer U, Michel P, Strambo D, Jovin TG, Raymond J, Zaidat OO, Ringleb PA, Nguyen TN, Nagel S. Reperfusion Without Functional Independence in Late Presentation of Stroke With Large Vessel Occlusion. Stroke. 2022 Dec;53(12):3594-3604. doi: 10.1161/STROKEAHA.122.039476. Epub 2022 Oct 14. PMID 36252092
- [Result] Siegler JE, Qureshi MM, Nogueira RG, Tanaka K, Nagel S, Michel P, Vigilante N, Ribo M, Yamagami H, Yoshimura S, Abdalkader M, Haussen DC, Mohammaden MH, Nannoni S, Mohlenbruch MA, Henon H, Sheth SA, Ortega-Gutierrez S, Olive-Gadea M, Caparros F, Seker F, Zaidi S, Castonguay AC, Uchida K, Sakai N, Puri AS, Farooqui M, Toyoda K, Salazar-Marioni S, Takeuchi M, Farzin B, Masoud HE, Kuhn AL, Rana A, Morimoto M, Shibata M, Nonaka T, Klein P, Sathya A, Kiley NL, Cordonnier C, Strambo D, Demeestere J, Ringleb PA, Roy D, Zaidat OO, Jovin TG, Kaesmacher J, Fischer U, Raymond J, Nguyen TN. Endovascular vs Medical Management for Late Anterior Large Vessel Occlusion With Prestroke Disability: Analysis of CLEAR and RESCUE-Japan. Neurology. 2023 Feb 14;100(7):e751-e763. doi: 10.1212/WNL.0000000000201543. Epub 2022 Nov 4. PMID 36332983
- [Result] Demeestere J, Qureshi MM, Vandewalle L, Wouters A, Strbian D, Nogueira RG, Nagel S, Yamagami H, Puetz V, Abdalkader M, Haussen DC, Mohammaden MH, Mohlenbruch MA, Olive-Gadea M, Winzer S, Ribo M, Michel P, Marto JP, Tanaka K, Yoshimura S, Martinez-Majander N, Caparros F, Henon H, Tomppo L, Dusart A, Bellante F, Ramos JN, Jesser J, Sheth SA, Ortega-Gutierrez S, Siegler JE, Nannoni S, Kaesmacher J, Dobrocky T, Salazar-Marioni S, Farooqui M, Virtanen P, Ventura R, Zaidi SF, Castonguay AC, Uchida K, Puri AS, Sakai N, Toyoda K, Farzin B, Masoud HE, Klein P, Bui J, Rizzo F, Kaiser DPO, Desfontaines P, Strambo D, Cordonnier C, Lin E, Ringleb PA, Roy D, Zaidat OO, Fischer U, Raymond J, Lemmens R, Nguyen TN. Outcomes of Bridging Intravenous Thrombolysis Versus Endovascular Therapy Alone in Late-Window Acute Ischemic Stroke. Stroke. 2024 Jul;55(7):1767-1775. doi: 10.1161/STROKEAHA.124.046495. Epub 2024 May 15. PMID 38748598
- [Result] Mujanovic A, Strbian D, Demeestere J, Marto JP, Puetz V, Nogueira RG, Abdalkader M, Nagel S, Raymond J, Ribo M, Michel P, Yoshimura S, Zaidat OO, Winzer S, Ortega-Gutierrez S, Sheth SA, Siegler JE, Dusart A, Haussen DC, Henon H, Serrallach BL, Mohammaden MH, Mohlenbruch MA, Olive-Gadea M, Puri AS, Sakai N, Klein P, Tomppo L, Caparros F, Ramos JN, Jumaa M, Zaidi S, Dobrocky T, Martinez-Majander N, Nannoni S, Bellante F, Rodriguez-Calienes A, Salazar-Marioni S, Virtanen P, Kaiser DP, Ventura R, Jesser J, Castonguay AC, Qureshi MM, Masoud HE, Galecio-Castillo M, Requena M, Lauha R, Hu W, Lin E, Miao Z, Roy D, Yamagami H, Seiffge DJ, Strambo D, Ringleb PA, Lemmens R, Fischer U, Nguyen TN, Kaesmacher J. Safety and clinical outcomes of endovascular therapy versus medical management in late presentation of large ischemic stroke. Eur Stroke J. 2024 Dec;9(4):907-917. doi: 10.1177/23969873241249406. Epub 2024 May 17. PMID 38757713
- [Result] Nguyen TN, Nogueira RG, Qureshi MM, Nagel S, Raymond J, Abdalkader M, Demeestere J, Marto JP, Sheth SA, Puetz V, Dusart A, Michel P, Ribo M, Zaidat OO, Siegler JE, Haussen DC, Strbian D, Henon H, Mohammaden MH, Mohlenbruch MA, Olive-Gadea M, Puri AS, Winzer S, Kaesmacher J, Klein P, Tomppo L, Caparros F, Ramos JN, Jumaa MA, Zaidi SF, Martinez-Majander N, Nannoni S, Vandewalle L, Bellante F, Farooqui M, Salazar-Marioni S, Virtanen P, Kaiser DPO, Wouters A, Ventura R, Jesser J, Mujanovic A, Shu L, Castonguay AC, Mansoor Z, Qiu Z, Masoud HE, Requena M, Peltola E, Hu W, Lin E, Tanaka K, Cordonnier C, Roy D, Yaghi S, Strambo D, Yamagami H, Fischer U, Jovin TG, Lemmens R, Ringleb PA, Ortega-Gutierrez S. Noncontrast CT Selected Thrombectomy vs Medical Management for Late-Window Anterior Large Vessel Occlusion. Neurology. 2024 May 28;102(10):e209324. doi: 10.1212/WNL.0000000000209324. Epub 2024 May 6. PMID 38709999
- [Result] Abdalkader M, Ning S, Qureshi MM, Haussen DC, Strbian D, Nagel S, Demeestere J, Puetz V, Mohammaden MH, Olive Gadea M, Winzer S, Yamagami H, Tanaka K, Marto JP, Tomppo L, Henon H, Sheth SA, Ortega-Gutierrez S, Martinez-Majander N, Caparros F, Lemmens R, Dusart A, Bellante F, Zaidi SF, Siegler JE, Nannoni S, Kaesmacher J, Dobrocky T, Farooqui M, Salazar-Marioni S, Virtanen P, Vandewalle L, Wouters A, Jesser J, Ventura R, Castonguay AC, Uchida K, Puri AS, Masoud HE, Klein P, Mansoor Z, Bui J, Kang M, Mujanovic A, Rizzo F, Kokkonen T, Ramos JN, Strambo D, Michel P, Mohlenbruch MA, Lin E, Kaiser DPO, Yoshimura S, Sakai N, Cordonnier C, Ringleb PA, Roy D, Zaidat OO, Fischer U, Ribo M, Raymond J, Nogueira RG, Nguyen TN. Sex Differences in Outcomes of Late-Window Endovascular Stroke Therapy. Stroke. 2024 Feb;55(2):278-287. doi: 10.1161/STROKEAHA.123.045015. Epub 2024 Jan 22. PMID 38252759
- [Derived] Tomppo L, Martinez-Majander N, Qureshi MM, Nguyen TN, Nogueira RG, Nagel S, Demeestere J, Puetz V, Henon H, Olive-Gadea M, Marto JP, Dusart A, Ringleb PA, Zaidat OO, Haussen DC, Mohammaden MH, Abdalkader M, Raymond J, Ortega-Gutierrez S, Sheth SA, Yamagami H, Ramos JN, Caparros F, Kaiser DPO, Ribo M, Salazar Marioni S, Tanaka K, Virtanen P, Puri AS, Siegler JE, Zaidi SF, Jumaa M, Lin E, Mayol J, Ventura R, Winzer S, Klein P, Bellante F, Cespedes J, Wouters A, Masoud HE, Shu L, Castonguay AC, Herweh C, Cheng M, Hu W, Roy D, Yaghi S, Lemmens R, Cordonnier C, Mohlenbruch MA, Strbian D. Outcomes of Witnessed Versus Unwitnessed Patients With Stroke After Endovascular Therapy in the Extended Time Window. Stroke. 2025 Nov 12. doi: 10.1161/STROKEAHA.125.052355. Online ahead of print. PMID 41221581
- [Derived] Winzer S, Kaiser DPO, Qureshi MM, Castonguay AC, Strbian D, Nogueira RG, Nagel S, Raymond J, Abdalkader M, Demeestere J, Marto JP, Yamagami H, Tanaka K, Sheth SA, Dusart A, Michel P, Olive Gadea M, Ribo M, Zaidat OO, Haussen DC, Henon H, Mohammaden MH, Mohlenbruch MA, Siegler JE, Puri AS, Kaesmacher J, Klein P, Tomppo L, Caparros F, Ramos JN, Jumaa M, Zaidi S, Martinez-Majander N, Nannoni S, Vandewalle L, Bellante F, Galecio-Castillo M, Salazar-Marioni S, Virtanen P, Wouters A, Ventura R, Jesser J, Mujanovic A, Shu L, Qureshi A, Qiu Z, Masoud HE, Requena M, Sillanpaa M, Hu W, Lin E, Cordonnier C, Roy D, Yaghi S, Strambo D, Fischer U, Ortega-Gutierrez S, Lemmens R, Ringleb PA, Nguyen TN, Puetz V. Endovascular Therapy for Late-Window M2-Segment Middle Cerebral Artery Occlusion: Analysis of the CLEAR Study. Stroke. 2025 Jul;56(7):1671-1680. doi: 10.1161/STROKEAHA.124.048840. Epub 2025 May 22. PMID 40405459
- [Derived] Marto JP, Qureshi M, Nagel S, Nogueira RG, Henon H, Tomppo L, Ringleb PA, Haussen DC, Abdalkader M, Puetz V, Zaidat OO, Demeestere J, Ramos JN, Ribo M, Olive-Gadea M, Mohammaden MH, Ortega-Gutierrez S, Sheth S, Yamagami H, Dusart A, Raymond J, Caparros F, Kaiser D, Tanaka K, Virtanen P, Puri AS, Siegler JE, Zaidi SF, Jumaa MA, Lin E, Requena M, Michel P, Winzer SM, Klein P, Nannoni S, Bellante F, Salazar-Marioni S, Galecio-Castillo M, Wouters A, Ventura R, Mujanovic A, Shu L, Castonguay AC, Jesser J, Masoud HE, Kaesmacher J, Hu W, Roy D, Yaghi S, Asdaghi N, Strambo D, Lemmens R, Strbian D, Cordonnier C, Mohlenbruch M, Nguyen TN. Endovascular Therapy for Patients With Low NIHSS Scores and Large Vessel Occlusion in the 6- to 24-Hour Window: Analysis of the CLEAR Study. Neurology. 2025 Apr;104(7):e213442. doi: 10.1212/WNL.0000000000213442. Epub 2025 Mar 20. PMID 40112237
- [Derived] Siegler JE, Koneru M, Qureshi MM, Doheim M, Nogueira RG, Martinez-Majander N, Nagel S, Penckofer M, Demeestere J, Puetz V, Ribo M, Abdalkader M, Marto JP, Al-Bayati AR, Yamagami H, Haussen DC, Olive-Gadea M, Winzer S, Mohammaden MH, Lemmens R, Tanaka K, Virtanen P, Dusart A, Bellante F, Kaiser DPO, Caparros F, Henon H, Ramos JN, Ortega-Gutierrez S, Sheth SA, Nannoni S, Vandewalle L, Kaesmacher J, Salazar-Marioni S, Tomppo L, Ventura R, Zaidi SF, Jumaa M, Castonguay AC, Galecio-Castillo M, Puri AS, Mujanovic A, Klein P, Shu L, Farzin B, Moomey H, Masoud HE, Jesser J, Mohlenbruch MA, Ringleb PA, Strbian D, Zaidat OO, Yaghi S, Strambo D, Michel P, Roy D, Yoshimura S, Uchida K, Raymond J, Nguyen TN. CLEAR Thrombectomy Score: An Index to Estimate the Probability of Good Functional Outcome With or Without Endovascular Treatment in the Late Window for Anterior Circulation Occlusion. J Am Heart Assoc. 2024 Jul 16;13(14):e034948. doi: 10.1161/JAHA.124.034948. Epub 2024 Jul 9. PMID 38979812
- See also: Endovascular Therapy in the Extended Time Window for Large Vessel Occlusion in Patients With Pre-Stroke Disability — https://j-stroke.org/journal/view.php?number=531